CLINICAL TRIAL: NCT04058873
Title: A Study on the Feasibility and Acceptability of Pericoital Levonorgestrel 1.5mg
Status: Completed | Type: Observational
Sponsor: Camber Collective (Other)
Collaborators: Population Council (Other); Marie Stopes International (Other); Bill and Melinda Gates Foundation (Other); The Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019LNG1.5mg
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

INTERVENTIONS:
Drug: Levonorgestrel 1.5mg — Levonorgestrel 1.5mg for pericoital use

SUMMARY:
This study intends to build on the previous research and gather data in an actual use study / patient registry of pericoital LNG 1.5mg to understand women's acceptability of the product along with associated side effects, and monitoring for their correct and incorrect use. These findings will contribute to the discussion around the feasibility of pericoital LNG as an additional contraceptive by adding to the body of evidence.

DETAILED DESCRIPTION:
The study would consist of distributing pericoital LNG 1.5mg across 75 pharmacy sites in Ghana over the course of 12 months. Recruitment will be staggered, and women will be recruited up to 9 months into the study. As such, the data collection period per participant will be at least 3 months.

Consistent with the recent WHO study (Festin et al. " A prospective, open-label, single arm, multicentre study to evaluate efficacy, safety and acceptability of pericoital oral contraception using LNG 1.5mg" (2016)), participants will be given instructions on how to correctly use LNG 1.5mg, namely to take one pill 24 hours before or after sexual relations, and no more than 6 times per month. Contraceptive protection requires use only once per 24 hours, regardless of how many times sexual relations are had during those 24 hours.

Participants will include a broad population of women age 18-49, not currently on any long-term modern method, who do not wish to get pregnant in the following 6 months but would not consider it a serious issue if they did become pregnant. They will be asked to use LNG 1.5mg as their exclusive method of contraception for the period of the study, with the exception of condoms.

The drug used for the study is LNG 1.5mg, specifically Marie Stopes International's BK-1 pill, repackaged for the study purposes. The BK-1 pill is currently registered as an emergency contraceptive and sold in Ghana with good quality assurance procedures in place. The BK-1 emergency contraception pill is manufactured for Marie Stopes International by Acme Formulation Pvt., Limited, one of the leading drug manufacturers of India. It is registered as an emergency contraception by the Food and Drugs Authority in Ghana and assigned registration number FDA/SD.183-11710. The package will read "LNG 1.5mg for Pericoital Use - for study purposes only" and be devoid of any other branding (please see Appendix for artwork).

Data collection components with research participants include:

1. Baseline background information about the research participants will be collected during the screening (e.g., qualifications for inclusion/ exclusion) and enrollment process
2. Biweekly (i.e., every two weeks) phone call surveys with research participants. They will be asked 10 questions about user satisfaction, circumstances of use, and outcomes (e.g., self-reported side effects)
3. Two extended surveys per participant to better understand participant perception of LNG 1.5mg, customer satisfaction with product and service, and future contraceptive intentions

Data collection components with pharmacies will include:

1. Baseline data of average packs of FP products sold at the pharmacy, in order to understand the overall increase in FP methods sold over the course of the study
2. A mystery shopping survey to check the quality of service provision and monitoring of recruitment/quality of information at each of the 75 study sites 2x during the study
3. Register collected at pharmacy point of sale, with units sold over the course of the 12-month pilot. Note: participants will be able to go to any of the participating pharmacies during the course of the project.
4. Pharmacists feedback surveys to understand the provision of LNG 1.5mg

ELIGIBILITY:
Inclusion Criteria:

* between the age of 18-49 years, is willing to use LNG 1.5 mg tablets as her primary contraceptive method, wants to avoid pregnancy for at least the next 6 months after enrollment, is willing to accept an uncertain risk of pregnancy during the study, and understands that the risk of pregnancy on this method would be slightly higher than other methods of contraception

Exclusion Criteria:

* women using one or more of the following contraceptive methods: daily pill, injectable, implant, sterilization

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female only
Study Population: women from areas surrounding distribution sites (pharmacies)
Sampling Method: Non-Probability Sample
Enrollment: 1980 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of use | 3-9 months
  Self reported via bi-weekly survey: women are able to access and use product correctly (consistent with instructions from health care provider / pharmacist)
Acceptability | 3-9 months
  Self reported via bi-weekly survey: Understand drivers behind decision-making of using pericoital LNG 1.5mg, conditions of use, and potential impact on increased mCPR and intention to use longer-term methods in the future

SECONDARY OUTCOMES:
Side effects | 3-9 months
  Self reported via bi-weekly survey: self reported side effects from using product

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Kuffour, Principal Investigator — AYA Collective
Locations (1):
- Marie Stopes International Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Festin MP, Bahamondes L, Nguyen TM, Habib N, Thamkhantho M, Singh K, Gosavi A, Bartfai G, Bito T, Bahamondes MV, Kapp N. A prospective, open-label, single arm, multicentre study to evaluate efficacy, safety and acceptability of pericoital oral contraception using levonorgestrel 1.5 mg. Hum Reprod. 2016 Mar;31(3):530-40. doi: 10.1093/humrep/dev341. Epub 2016 Jan 31. PMID 26830816